CLINICAL TRIAL: NCT05235568
Title: Prospective, Single-arm Pivotal Study for the Treatment of Subjects With Severe Symptomatic Calcific Aortic Valve Stenosis Using Valvosoft® Non-Invasive Ultrasound Therapy (NIUT)
Brief Title: VALVOSOFT® Pivotal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiawave SA (Industry)
Collaborators: QbD Clinical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CW21-02
Record Dates: First submitted 2022-01-20; First posted 2022-02-11 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Aortic Valve Calcification; Aortic Valve Stenosis
Keywords: Aortic Valve Stenosis; Aortic Valve Calcification; Aortic Valve; Stenosis; Ultrasound; non invasive
MeSH Terms: conditions — Aortic Valve, Calcification of; Aortic Valve Stenosis; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Valvosoft (Other): Treatment with VALVOSOFT device
  Interventions: Device: VALVOSFT intervention

INTERVENTIONS:
Device: VALVOSFT intervention — Treatment of the calcific aorta valve by non-invasive ultrasound therapy

SUMMARY:
The objective of the study is to evaluate the safety and performance of a new non-invasive ultrasound therapy (NIUT) with Valvosoft in the treatment of Calified Aortic Stenosis

ELIGIBILITY:
Inclusion Criteria:

1. Subject suffering from severe symptomatic calcific aortic valve stenosis as defined by ESC/EACTS guidelines for the management of valvular heart disease 2021; and
2. Subject is not recommended by the local HEART Team for immediate TAVR/SAVR; or
3. Subject who refuses TAVR/SAVR, documented by local HEART Team (not allowed in France); and
4. Age ≥18 years; and
5. Subject willing to provide a written informed consent prior to participating in the study; and
6. Subject who can comply with the study follow-up or other study requirements; and
7. Subject is eligible for the Valvosoft procedure according to Clinical Review Committee (CRC).

Exclusion Criteria:

1. Subject with severe aortic regurgitation; or
2. Subject with unstable arrhythmia not controlled by medical treatment; or
3. Subjects with implanted mechanical valve in any position or bio-prosthetic valve in aortic position; or
4. Subject has a chest deformity not allowing optimal placement of Valvosoft Applicator and visualization of the aortic valve; or
5. Cardiogenic shock or other hemodynamic instability; or
6. Left Ventricular Ejection Fraction ≤30%; or
7. Subject with mean AVAI <0,24 cm²/m2; or
8. History of heart transplant; or
9. Subject requiring other cardiac surgery procedures (bypass graft surgery, mitral valve procedure, tricuspid valve procedure) within one month after Valvosoft procedure; or
10. Cardiac imaging evidence of vegetation; or
11. Acute myocardial infarction (MI) within one month prior to enrolment; or
12. Valve depth not suitable for NIUT (depth >125mm with respect to the Valvosoft imaging probe); or
13. Stroke or transient ischemic attack (TIA) ≤1 month prior to enrollment; or
14. Subject who is pregnant, or plan to become pregnant during the 12-months study follow-up period; or
15. Subject who is participating in another research study for which the primary endpoint has not been reached; or
16. Balloon aortic valvuloplasty (BAV) ≤3 months prior to enrollment; or
17. Current endocarditis; or
18. Leukopenia (WBC <4000 cell/μL), anemia (Hgb <8 g/dL), thrombocytopenia (platelet count <15.000 cell/μL), or history of coagulopathy or hypercoagulable state; or
19. Life expectancy < 6 months due to non-cardiac co-morbid conditions; or
20. Other medical, psychological, or social condition which, in the opinion of the investigator, precludes the subject from study participation; or
21. Subjects who do not have Social Security and who are under legal restraint; or
22. Subjects who cannot read or write or are mentally not or partially capable of giving informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Safety endpoint | at 30 days post-procedure
  Rate of MACE < 25%
Performance endpoint | at 30 days post-procedure
  Improvement in clinical status assessed by means of a decrease in NHYA functional class

SECONDARY OUTCOMES:
Rate of MACE | peri-procedureal, and at 3-, 6- and 12 months post procedure
  Rate of major adverse and cerebral events
All cause mortality | 30 days, 3-, 6- and 12-months post procedure
  All cause mortality
Rate of Stroke | 30 days, 3-, 6- and 12-months post procedure;
  Rate of stroke (disabling and non-disabling; ischemic and hemorrhagic)
AVA change at 30 days | 30 days post procedure
  Change of 10% in of aortic stenosis by means of aortic valve area (AVA) (assessed by the independent echocardiographic Central Core Laboratory) 30 days post procedure compared to baseline
AVA change in severity | at 6- and 12 months
  Change in severity of aortic stenosis by means of aortic valve area (AVA) (assessed by the independent echocardiographic Central Core Laboratory) at 6- and 12 months compared to baseline
NYHA improvement | 3-, 6- and 12-months
  Change in clinical status assessed by means of a decrease in NYHA functional class
Change in 6 minutes walk test | 30 days, 6- and 12 months
  Change in 6-minutes' walk test
Improvement of quality of life by Kansas City Cardiomyopathy Questionnaire (KCCQ) | 30 days, 6-, and 12-months
  Improvement of quality of life by means of KCCQ. KCCQ is a 23-item, self-administered questionnaire
Improvement of quality of life by EQ-5D | 30 days, 6-, and 12-months
  Improvement of quality of life by means of EQ-5D. The EQ-5D descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Spaulding, MD, PhD, Principal Investigator — HEGP, Paris, France
Locations (11):
- France (6):
  - CHU Lille Insitut Coeur Poumon, Lille
  - Hopital Bichat Claude-Bernard, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - CHU Reims Hopital Robert Debré, Reims
  - CHU Rouen Hopital Charles Nicole, Rouen
  - Clinique Pasteur, Toulouse
- Germany (2):
  - Kerckhoff-klinik, Bad Nauheim
  - Marienkrankenhaus, Hamburg
- Netherlands (3):
  - OLVG, Amsterdam
  - Amphia Hospital, Breda
  - Radboudumc, Nijmegen

IPD SHARING:
Plan to Share IPD: No